CLINICAL TRIAL: NCT05107726
Title: Piloting a Family-Based Intervention of Time-Restricted Eating to Treat Obesity
Brief Title: Family Based Time-Restricted Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2021-30078
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: A total of 20 dyads will be enrolled in this study. A dyad will consist of a parent and a child. Dyads will be randomized to one of two treatment groups: the time restricted eating (TRE) group or standard of care control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRE Group (Experimental): In the TRE group, study staff will instruct the family unit on limiting the eating window to 10-12 hours per day, during which they can eat ad libitum. Notably, in the TRE group, participants (children and adults) will be instructed to brush their teeth with a WIFI-enabled toothbrush in the morning and specifically within ½ hour after their evening meal. This will serve as a cue to stop evening eating, and information from the WIFI-enabled toothbrush will be accessed by study staff to approximate the eating window. The adult from each family unit will receive a daily REDCap-administered email to indicate the timing of the first meal of the day and the last meal of the day for the parent and child, which will also serve as an estimate of the eating window.
  Interventions: Behavioral: TRE Group
- Standard of Care Group (No Intervention): The standard of care control group will receive dietary instruction that is based on a 1200-1500 calorie diet, as is typical of family-based interventions. Calorie counting will not be encouraged. However, families will be encouraged to follow appropriate portion sizes; increase vegetable, fruit and lean protein consumption; as well as decrease consumption of energy-dense but low-quality items (e.g., sugar sweetened beverages). Families in this group will also receive a WIFI-enabled toothbrush and daily REDCap surveys but will not be instructed on when to brush teeth or to shorten their eating window

INTERVENTIONS:
Behavioral: TRE Group — This group will practice time-restricted eating
  Arms: TRE Group

SUMMARY:
This study will test whether managing the hours during which people eat, called time restricted eating, might help them to lose weight. For this study, one parent and a child will enroll as a group (called a dyad).

The dyads will be assigned at random to practice time restricted eating (within 10-12 hours per day) but will be able to eat whatever they would like or to limit portion size and increase fruit, vegetable and lean protein intake and limit sugar sweetened beverages and undergo . Both groups will receive dietary counseling, Bluetooth toothbrushes and scales to help monitor their progress.

The study will last for 12 weeks and will have one survey four weeks after the last in person visit. There will be 2 in person visits, 7 virtual visits, 2 phone visits and daily time logs.

DETAILED DESCRIPTION:
This study will provide preliminary data to demonstrate feasibility and acceptability of time-restricted eating (TRE) in the family unit, providing critical preliminary data to support NIH-level funding for a more detailed analysis of TRE in families.

Obesity affects over 40% of adults and over 25% of children in the United States. Obesity - defined in adults as a body mass index (BMI) > 30 kg/m2 and in children as BMI > 95th percentile - is associated with several physical and psychological comorbidities, such as hypertension, heart disease, type 2 diabetes mellitus, and reduced quality of life. Heritability of obesity is 40-75%. Thus, if a parent is obese, children in the family have a high likelihood of also becoming obese due to both genetic and environmental factors. As such, treatments that apply to the family unit can address the public health concern of obesity at the child and adult level.

Typically, obesity treatment primarily focuses on intentional caloric restriction. In adults with obesity, behavior-based weight loss programs result in weight reduction of 1-4 kg over one year. In children with obesity, lifestyle modification therapy typically results in weight stabilization, while children without treatment gain weight. Weight stabilization results in reductions in body mass index parameters (e.g., percent BMI or BMI z-score) due to increased height in children. Family-based obesity treatment also focuses on intentional caloric restriction through reduced consumption of energy dense foods, as well as increased consumption of low energy density foods, increased physical activity, and implementation of strategic parenting practices. Parent BMI change is a significant predictor of child outcomes in family-based treatment. Unfortunately, family-based interventions are typically time and resource intensive, thus limiting their receptiveness by many families.

In contrast to intentionally restricting calories, time-restricted eating (TRE) intentionally restricts the eating window while allowing ad libitum intake during the window. TRE's agnostic approach to eating allows individuals to select foods that align with their needs and preferences. Multiple studies in adults, including our own, demonstrate TRE reduces weight. The postulated mechanism is that a reduced eating window reduces the number of eating occasions to reduce daily caloric intake.

ELIGIBILITY:
Inclusion Criteria:

* BMI >/= 30 kg/m2 for the parent
* BMI > 95th percentile for the child
* Age 3-9 years for the child
* Age >/= 18 years old for the parent

Exclusion Criteria:

* Concurrent participation in another weight loss study
* Taking any medications for weight loss
* Pregnancy or anticipation of pregnancy in next 6 months (for the parent)
* 3+ on Eating Disorder Survey

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | 12 weeks
  Change in body mass index from Screening to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Amy Gross, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Delaware Clinical Research Unit, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT05107726/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT05107726/ICF_001.pdf